CLINICAL TRIAL: NCT01139515
Title: An Open Label, Single And Repeat Dose Randomized Crossover Study To Estimate The Pharmacokinetics And Safety Of Eletriptan Hydrobromide Tablets In Healthy Korean Male Subjects
Brief Title: Eletriptan Pharmacokinetics In Korean Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1601126
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: pharmacokinetic; eletriptan; Korean; crossover

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): 1 X 20 mg eletriptan
  Interventions: Drug: Eletriptan commercial tablet
- Treatment B (Experimental): 1 X 40 mg eletriptan
  Interventions: Drug: Eletriptan commercial tablet
- Treatment C (Experimental): 2 X 40 mg eletriptan
  Interventions: Drug: Eletriptan commercial tablet
- Treatment D (Experimental): 1 X 40 mg tablet given 2 hr after initial 1 X 40 mg tablet dose
  Interventions: Drug: Eletriptan commercial tablet

INTERVENTIONS:
Drug: Eletriptan commercial tablet — 20 mg tablet, single dose
  Arms: Treatment A
Drug: Eletriptan commercial tablet — 40 mg tablet, single dose of 1 X 40 mg
  Arms: Treatment B
Drug: Eletriptan commercial tablet — 40 mg tablet, single dose of 2 X 40 mg
  Arms: Treatment C
Drug: Eletriptan commercial tablet — 40 mg tablet, 1 X 40 mg given two times: the second 2 hours after the first
  Arms: Treatment D

SUMMARY:
The hypothesis of this study is that Korean subjects have similar Pharmacokinetics (PK) characteristics to those seen in other populations.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects, 18-55 years old
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2
* provide informed consent

Exclusion Criteria:

* blood pressure >140/90 mm Hg
* any condition possibly affecting drug absorption
* positive urine drug screen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1601126&StudyName=Eletriptan%20Pharmacokinetics%20In%20Korean%20Males

RESULTS

PARTICIPANT FLOW:
Groups:
- Eletriptan 20 mg,40 mg,80 mg,40 mg 2 Hrs Apart Repeated Dose: Single oral dose of eletriptan 20 mg tablet in first intervention period; followed by single oral dose of eletriptan 40 mg tablet in second intervention period; then single oral dose of eletriptan 80 mg tablet in third intervention period; and two oral doses of 40 mg eletriptan tablet administered 2 hrs apart in fourth intervention period. A washout period of 46 hrs was maintained between each period.
- Eletriptan 40 mg,80 mg,20 mg,40 mg 2 Hrs Apart Repeated Dose: Single oral dose of eletriptan 40 mg tablet in first intervention period; followed by single oral dose of eletriptan 80 mg tablet in second intervention period; then single oral dose of eletriptan 20 mg tablet in third intervention period; and two oral doses of 40 mg eletriptan tablet administered 2 hrs apart in fourth intervention period. A washout period of 46 hrs was maintained between each period.
- Eletriptan 80 mg,40 mg 2 Hrs Apart Repeated Dose,40 mg,20 mg: Single oral dose of eletriptan 80 mg tablet in first intervention period; followed by two oral doses of 40 mg eletriptan tablet administered 2 hrs apart in second intervention period; then single oral dose of eletriptan 40 mg tablet in third intervention period; and single oral dose of eletriptan 20 mg tablet in fourth intervention period. A washout period of 46 hrs was maintained between each period.
- Eletriptan 40 mg 2 Hrs Apart Repeated Dose,20 mg,80 mg,40 mg: Two oral doses of 40 mg eletriptan tablet administered 2 hrs apart tablet in first intervention period; followed by single oral dose of eletriptan 20 mg in second intervention period; then single oral dose of eletriptan 80 mg tablet in third intervention period; and single oral dose of eletriptan 40 mg tablet in fourth intervention period. A washout period of 46 hrs was maintained between each period.
Period: First Intervention Period
Arm/Group | Eletriptan 20 mg,40 mg,80 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 40 mg,80 mg,20 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 80 mg,40 mg 2 Hrs Apart Repeated Dose,40 mg,20 mg | Eletriptan 40 mg 2 Hrs Apart Repeated Dose,20 mg,80 mg,40 mg
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period I (46hrs)
Arm/Group | Eletriptan 20 mg,40 mg,80 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 40 mg,80 mg,20 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 80 mg,40 mg 2 Hrs Apart Repeated Dose,40 mg,20 mg | Eletriptan 40 mg 2 Hrs Apart Repeated Dose,20 mg,80 mg,40 mg
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Eletriptan 20 mg,40 mg,80 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 40 mg,80 mg,20 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 80 mg,40 mg 2 Hrs Apart Repeated Dose,40 mg,20 mg | Eletriptan 40 mg 2 Hrs Apart Repeated Dose,20 mg,80 mg,40 mg
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (46 Hrs)
Arm/Group | Eletriptan 20 mg,40 mg,80 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 40 mg,80 mg,20 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 80 mg,40 mg 2 Hrs Apart Repeated Dose,40 mg,20 mg | Eletriptan 40 mg 2 Hrs Apart Repeated Dose,20 mg,80 mg,40 mg
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Eletriptan 20 mg,40 mg,80 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 40 mg,80 mg,20 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 80 mg,40 mg 2 Hrs Apart Repeated Dose,40 mg,20 mg | Eletriptan 40 mg 2 Hrs Apart Repeated Dose,20 mg,80 mg,40 mg
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3 (46 Hrs)
Arm/Group | Eletriptan 20 mg,40 mg,80 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 40 mg,80 mg,20 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 80 mg,40 mg 2 Hrs Apart Repeated Dose,40 mg,20 mg | Eletriptan 40 mg 2 Hrs Apart Repeated Dose,20 mg,80 mg,40 mg
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | Eletriptan 20 mg,40 mg,80 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 40 mg,80 mg,20 mg,40 mg 2 Hrs Apart Repeated Dose | Eletriptan 80 mg,40 mg 2 Hrs Apart Repeated Dose,40 mg,20 mg | Eletriptan 40 mg 2 Hrs Apart Repeated Dose,20 mg,80 mg,40 mg
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All participants randomized to any treatment (Eletriptan 20 mg tablet first, eletriptan 40 mg tablet first, eletriptan 80 mg tablet first, and eletriptan 40 mg 2 hrs apart repeated dose (80 mg in total).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)]
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: Pre-dosing, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hrs post dose (A,B,C) and additional 2.5,2.75,3.5,5,14,18 and 26 hrs post dose(D)
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Full Range); unit: ng* hr/mL
Groups:
- Eletriptan 20 mg Tablet: Single oral dose of eletriptan 20 mg tablet (Treatment A).
- Eletriptan 40 mg Tablet: Single oral dose of eletriptan 40 mg tablet (Treatment B).
- Eletriptan 80 mg Tablet: Single oral dose of two eletriptan 40 mg tablets (Treatment C).
- Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose: Repeated oral dose of eletriptan 40 mg tablet administered 2 hrs apart (total dose = 80 mg). (Treatment D).
Arm/Group | Eletriptan 20 mg Tablet | Eletriptan 40 mg Tablet | Eletriptan 80 mg Tablet | Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng* hr/mL | 291.3 [185.0 to 690.0] | 575.6 [358.0 to 1230.0] | 1282.0 [806.0 to 2140.0] | 1278.0 [842.0 to 2310.0]
Statistical Analysis 1: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 40 mg Tablet; Natural log transformed, dose-normalized AUC[0- ∞] of eletriptan was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect.The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Adjusted ratio of geometric means = 98.70, 90% CI 2-sided [92.17 to 105.70]
Statistical Analysis 2: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted ratio of geometric means = 109.48, 90% CI 2-sided [102.23 to 117.24]
Statistical Analysis 3: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 80 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted ratio of geometric means = 109.93, 90% CI 2-sided [102.65 to 117.72]

2. Primary Outcome: AUC From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration-time curve from time zero (pre-dose) to the time of the last measurable concentration (AUClast).
Time Frame: Pre-dosing, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hrs post dose (A,B,C) and additional 2.5,2.75,3.5,5,14,18 and 26 hrs post dose (D)
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Full Range); unit: ng*hr/mL
Arm/Group | Eletriptan 20 mg Tablet | Eletriptan 40 mg Tablet | Eletriptan 80 mg Tablet | Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng*hr/mL | 281.2 [180.0 to 646.0] | 558.7 [351.0 to 1160.0] | 1243.0 [767.0 to 2080.0] | 1244.0 [808.0 to 2210.0]
Statistical Analysis 1: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 40 mg Tablet; Natural log transformed, dose-normalized AUClast of eletriptan was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect.The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Adjusted geometric means ratio = 99.41, 90% CI 2-sided [92.97 to 106.31]
Statistical Analysis 2: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Adjusted ratio of geometric means = 110.52, 90% CI 2-sided [103.36 to 118.18]
Statistical Analysis 3: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 80 mg Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Adjusted ratio of geometric means = 110.44, 90% CI 2-sided [103.28 to 118.09]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Eletriptan 20 mg Tablet | Eletriptan 40 mg Tablet | Eletriptan 80 mg Tablet | Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 46.50 [29.50 to 97.80] | 94.72 [47.50 to 224.00] | 200.10 [77.80 to 423.00] | 183.60 [97.00 to 281.00]
Statistical Analysis 1: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 40 mg Tablet; Natural log transformed, dose-normalized Cmax of eletriptan was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Adjusted geometric means ratio = 101.81, 90% CI 2-sided [85.97 to 120.58]
Statistical Analysis 2: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Adjusted ratio of geometric means = 98.57, 90% CI 2-sided [83.23 to 116.73]
Statistical Analysis 3: Comparison: Eletriptan 20 mg Tablet vs Eletriptan 80 mg Tablet; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Adjusted ratio of geometric means = 107.44, 90% CI 2-sided [90.72 to 127.25]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hr
Arm/Group | Eletriptan 20 mg Tablet | Eletriptan 40 mg Tablet | Eletriptan 80 mg Tablet | Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose
Number analyzed (Participants) | 16 | 16 | 16 | 16
Hr | 0.750 [0.500 to 2.000] | 0.750 [0.500 to 4.000] | 0.750 [0.500 to 6.000] | 5.000 [0.750 to 5.020]

5. Secondary Outcome: Plasma Decay Half Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hr
Arm/Group | Eletriptan 20 mg Tablet | Eletriptan 40 mg Tablet | Eletriptan 80 mg Tablet | Eletriptan 40 mg Tablet 2 Hrs Apart Repeated Dose
Number analyzed (Participants) | 16 | 16 | 16 | 16
Hr | 4.924 (0.685) | 4.630 (0.447) | 4.576 (0.531) | 4.753 (0.623)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Eletriptan 40 mg 2 Hrs Apart Repeated Dose: Repeated oral dose of eletriptan 40 mg tablet administered 2 hrs apart (total dose = 80 mg). (Treatment D).
Arm/Group | Eletriptan 20 mg Tablet | Eletriptan 40 mg Tablet | Eletriptan 80 mg Tablet | Eletriptan 40 mg 2 Hrs Apart Repeated Dose
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16 | 4/16 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eletriptan 20 mg Tablet (N=16) | Eletriptan 40 mg Tablet (N=16) | Eletriptan 80 mg Tablet (N=16) | Eletriptan 40 mg 2 Hrs Apart Repeated Dose (N=16)
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Oral mucosa erosion (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.